CLINICAL TRIAL: NCT00164229
Title: Study to Investigate the Effectiveness of a Math Intervention for Children With Fetal Alcohol Syndrome or Related Condition
Brief Title: Fetal Alcohol Syndrome: Socio-Cognitive Habilitation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Emory University (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Marcus Institute (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CDC-NCBDDD-3721; U84ccu320162
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2005-09

CONDITIONS: Fetal Alcohol Syndrome
Keywords: treatment; control
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

INTERVENTIONS:
Behavioral: math
Behavioral: behavior regulation

SUMMARY:
Comprehensive evaluation (geneticist, psychologist, social worker, education specialist, others as indicated) to determine individual needs and treatment plan. Referrals for specific services (e.g., OT, counseling, medications, etc) will be to clinicians within the families' own communities. All families will receive evaluation, parent education/advocacy, and learning readiness program. Only the intervention group will receive the math intervention.

DETAILED DESCRIPTION:
Learning Readiness Program: This program will include: case management to secure needed services, medication consultation (psychiatrist), educational consultation/ liaison, Behavioral Regulation Training (BRT). BRT will include teaching parents about: 1) recognizing their child's arousal level (to avoid negative episodes), 2) recognizing their own arousal and how it contributes to a situation, 3) principles of social reinforcement (e.g., praise, ignore, etc), 4) "accidental teaching" (i.e., teaching when a situation/opportunity arises), 5) resource/support source identification, 6) to communicate choices rather than authoritative commands, and 6) reduction of repetitive prompts (nagging). The child will be taught: 1) the technique of Escape/No Escape for undesirable tasks, 2) arousal awareness, and 3) verbalization of situations and actions (e.g., I don't like it when mom yells at me for running in the house, so I won't run in the house).

Targeted Area of Intervention: MATH - 6 weeks of individualized math tutoring. Content of the tutoring will be tailored to age levels (either 3-6 yr olds or 6-9 yr olds). The High/Scope curriculum will be used (modified so that it can be individualized). In addition, visual materials and visual aids will be developed to address deficits in the visual-spatial skills of children with FAS/ARND. For teachers, a manual will be prepared to assist them in working with children who have FAS/ARND. The educational specialist will review the manual and techniques with each teacher involved with the child.

Parent component: Individual and small group sessions to include: FAS education, information on education system procedures, instruction for communicating with professionals, and support for advocating for their child. A caregiver manual will be prepared.

Evaluation Plan: Treatment and control groups will be compared using pre- and post-tests measures. Post-tests will be at the conclusion of the intervention and at a 6-month follow-up. Process (e.g., parent satisfaction, compliance, etc) and outcome (e.g., math skill, behavior, family functioning, etc) measures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of FAS or related condition
* age 3 years six month or older

Exclusion Criteria:

* age 6 years 9 months or older

Ages: 42 Months to 81 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2001-10; Study Completion 2005-01

PRIMARY OUTCOMES:
math knowledge
math skills

SECONDARY OUTCOMES:
behavior regulation
parent knowledge of FAS

CONTACTS AND LOCATIONS:
Overall Officials: claire coles, PhD, Principal Investigator — Marcus Institute
Locations (1):
- Marcus Institute, Atlanta, Georgia, United States